CLINICAL TRIAL: NCT02877108
Title: An Observational Study of Anti-Psychotic Medication for the Treatment of Agitation in the Emergency Department
Brief Title: Naturalistic Adasuve Clinical Trial Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mt Sinai Hospital, Chicago (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Leslie Zun, MD, Chairman of Emergency Department, Mt Sinai Hospital, Chicago
Other Study IDs: 15-26
Record Dates: First submitted 2015-08-20; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adasuve: These patients will receive Adasuve for treatment of agitation.
- Haloperidol/Lorazepam: These patients will receive haloperidol/lorazepam for treatment of agitation.

SUMMARY:
There is limited information on the best psychoactive medication to treat agitated patients in the emergency department. The intent of this study is to fill in knowledge gaps in the current practice of treating psychiatric patients in the acute care setting. The purpose of this study is to determine the best treatment for agitated psychiatric patients in the emergency department.

DETAILED DESCRIPTION:
Patients with psychiatric complaints frequently present for evaluation and treatment in emergency departments across the country. In particular, agitation in the emergency department can have life-threatening consequences for both patients and staff, and so patients are frequently given medications to reduce their level of agitation and permit medical examination.

Primary and secondary objectives:

The primary objective of this study is to compare the efficacy and effectiveness of inhaled loxapine (Adasuve) vs. traditional emergency department treatment with intramuscular haloperidol with and without lorazepam in patients who present to the emergency department in an acutely agitated state. The Positive and Negative Syndrome Scale (PANSS-EC), Agitation and Calmness Evaluation Scale (ACES) will be used as measurements of agitation and Barnes akathisia scale will be used as measurements of side effects.

There are five secondary objectives: (1) To assess the level of agitation of psychiatric patients presenting to the emergency department using the PANSS-EC, ACES and Barnes scale; (2) To determine the effect of the level of agitation related to medication treatment and physical restraint using the PANSS-EC; (3) To determine the complication rate of the various medications administered with and without physical restraint; (4) To compare the effectiveness of various pharmacologic agents used in the emergency department for agitation using the delta of agitation over time (5) To determine the effect of the treatment choice on emergency department throughout time using emergency department (ED) throughput time.

Hypothesis:

The hypothesis of this study is to demonstrate superiority of inhaled loxapine (Adasuve) to the traditional anti-psychotic agents (with or without benzodiazepine) in the effectiveness of the treatment of agitation at 15 minute treatment time.

Research design:

The study is an observational convenience (when a research assistant is available), analysis of patients who are given psychoactive medications in the emergency department for agitation during a twelve month period.

The study will determine the level of patient agitation using the Positive and Negative Syndrome Scale (PANSS-EC), Agitation and Calmness Evaluation Scale (ACES) and Barnes akathisia scale. These scales were chosen because of their usage and applicability in studies of the treatment of agitation. The scales will be administered to the patients upon arrival, at fifteen minutes for the first hour and then every half hour for the next 2.5 hours or until the patient leaves the emergency department. The time medications are administered will be documented.

All agitated patients presenting to Mount Sinai Hospital emergency departments who, in the judgment of an ED clinician require treatment. Patients will be treated within the standard of care with the additional of one additional FDA approved medication. All agitated patients presenting to the ED with a psychiatric related complaint, in the judgement of the ED clinician will be prescribed a treatment of choice. The choices will include inhaled loxapine (Adasuve) vs. traditional emergency department treatment with intramuscular haloperidol with and without lorazepam. Clinicians will be free to prescribe any medication that they feel benefits the patient.

Research associates will approach patients who the emergency physician has deemed as agitated and in need of treatment. The research associate will obtain consent from the patient or their surrogate, if patient is not competent to consent to use the patient's information and ensure that the patient meets all study inclusion and no exclusion criteria. If the patient does not have the capacity to consent and no surrogate is available to consent, we will obtain patient data. When the patient gains capacity to consent, they will be approached to consent for use of their information that is being captured. Should these patients refuse consent; all information obtained will be destroyed.

The research associate will obtain consent from the patient or their surrogate and ensure that the patient meets all study inclusion and no exclusion criteria. The researcher will observe the patient and record the level of agitation over a 2.5 hour time period. The research associate will complete all study documents.

All patients will be evaluated by the emergency physician to provide medical clearance. The primary purpose of medical clearance is to determine whether a medical illness is causing or exacerbating the psychiatric condition. The secondary purpose is to identify medical or surgical conditions incidental to the psychiatric problem that may need treatment. The emergency service is responsible for the evaluation and treatment of a patients' agitation. They will determine the need for and choice of treatment option for the patient.

Teva Pharmaceuticals will provide a supply of Loxapine (Adasuve) for the emergency department for the time period of the study. The Principle Investigator has been in communication with the Pharmacy department regarding the storage and distribution of the drug. Please see inclusion/exclusion criteria in "Eligibility". The emergency department staff will be educated about the appropriate use of this education.

The research associate will obtain all necessary data elements either from the patient or the medical record. They will observe and record the PANSS-EC, ACES, and Barnes scores on each enrolled patient every fifteen minutes for the first hour then every half hour for a total of 2.5 hours or until the patient leaves the emergency department. Information will be collected on a data collection sheet that will include basic demographic information on the patient, age, gender, diagnosis, current medication, level of agitation before and after treatment, number of restraints, vital signs, time restraints were applied, type and time medication is administered and complications of therapy. A research associate will complete the data collection sheet and input the data of enrolled patients. The patients' psychiatric diagnosis from the psychiatric service will be noted. The research fellow will complete all study documents. The statistician will perform an analysis of the data looking for statistical significance of the data to the posed questions. Once all data is collected, any identifying information on the patient will be destroyed to ensure patient confidentiality.

Following data collection, the data will be analyzed using commercially-available software packages (such SPSS) to determine agitation reduction using 95% confidence intervals to exclude the margin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years of age and less than 65 years of age
* Patients must be emergency department patients during time of study
* All patients will be evaluated by the emergency physician to provide medical clearance- patients must be considered by the emergency physicians to be clinically agitated and to be clinically appropriate candidates for treatment with a medication
* Each patient, or a surrogate, must understand the nature of the study and must sign an informed consent document
* English speaking patients

Exclusion Criteria:

* Female patients who are either pregnant or breast-feeding
* Medically unstable patients
* Patients who have delirium or dementia
* Prisoners
* Patients <18 or >65 years old
* Non-English speaking patients
* Contraindications for use for people with asthma, COPD, and other acute respiratory conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department who are or become agitated, requiring medication
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Reduction of Agitation as Measured by the PANSS-CC | Three Hours
  Patients will receive either an inhaled loxapine or the traditional treatment of haloperidol and will be observed over a three hour period to compare effectiveness of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Zun, MD, Study Director — Sinai Health System
Locations (2):
- United States (2):
  - UCSD, La Jolla, California
  - Mount Sinai Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish findings once data enrollment and data analysis is complete.

REFERENCES:
- [Derived] Cole JB, Klein LR, Mullinax SZ, Nordstrom KD, Driver BE, Wilson MP. Study Enrollment When "Preconsent" Is Utilized for a Randomized Clinical Trial of Two Treatments for Acute Agitation in the Emergency Department. Acad Emerg Med. 2019 May;26(5):559-566. doi: 10.1111/acem.13673. Epub 2019 Jan 15. PMID 30548977